CLINICAL TRIAL: NCT02361333
Title: Barriers to Use of Remote Monitoring in Patients With Implantable Cardioverter Defibrillators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1208010730
Record Dates: First submitted 2015-01-20; First posted 2015-02-11 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Cardiac Patients; Implantable Cardioverter Defibrillator

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teaching Intervention (Experimental): Patients will be taught how to install and use a remote monitor.
  Interventions: Behavioral: Teaching Intervention
- No Intervention (No Intervention): Patients will not be taught how to install and use a remote monitor

INTERVENTIONS:
Behavioral: Teaching Intervention — Patients will be taught how to install and use a remote monitor
  Arms: Teaching Intervention

SUMMARY:
The purpose of this study is to determine whether a teaching intervention can help increase the use of remote monitors in patients with implantable cardioverter defibrillators.

ELIGIBILITY:
Inclusion Criteria:

* Received a Medtronic implantable cardioverter defibrillator (ICD) at Yale Electrophysiology, between January 2007 and June 2012
* ICD is compatible with Carelink, Medtronic's remote monitoring system

Exclusion Criteria:

* Less than 18 years of age
* From a vulnerable population
* Incompetent/suffers from dementia
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Number of remote Transmissions of data using remote monitor made by patient | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Yale Electrophysiology, New Haven, Connecticut, United States